CLINICAL TRIAL: NCT03196791
Title: A Double-blind, Randomized and Controlled Multicenter Prospective Trial to Compare the Oncological Benefit of Deep Neuromuscular Block in Gastric Cancer Obesity Patient
Brief Title: Compare the Oncological Benefit of Deep Neuromuscular Block in Gastric Cancer Obesity Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Debloqs_GC
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer; Obesity
MeSH Terms: conditions — Stomach Neoplasms; Obesity | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular block group (Experimental): Sugammadex sodium 4mg/kg/IV after operation
  Interventions: Drug: Sugammadex Sodium
- Moderate neuromuscular group (Experimental): Sugammadex sodium 2mg/kg/IV after operation
  Interventions: Drug: Sugammadex Sodium

INTERVENTIONS:
Drug: Sugammadex Sodium — 1. INDICATIONS AND USAGE BRIDION® is indicated for the reversal of neuromuscular blockade induced by rocuronium bromide and vecuronium bromide in adults undergoing surgery. BRIDION (sugammadex) injection is a sterile, clear, colorless to slightly yellow-brown, non-pyrogenic aqueous solution intended for intravenous infusion.
  2. DOSAGE AND ADMINISTRATION BRIDION (sugammadex) injection, for intravenous use, should be administered by trained healthcare providers familiar with the use, actions, characteristics, and complications of neuromuscular blocking agents (NMBA) and neuromuscular block reversal agents.
  Other Names: Bridion®, MSD

SUMMARY:
This study is designed to evaluate the impact of muscle relaxation during laparoscopic gastrectomy on oncological benefit, especially with obese patients over BMI 25. The primary endpoint is number of harvested lymph node that is critical point regarding quality of surgery in gastric cancer treatment. The secondary endpoint is intraoperative bleeding, surgeons' satisfaction.

The patients were randomly assigned to two groups using a computer-generated randomization table : 196 persons

* Deep neuromuscular block group (98persons)
* Moderate neuromuscular group (98persons)

DETAILED DESCRIPTION:
This study is designed to evaluate the impact of muscle relaxation during laparoscopic gastrectomy on oncological benefit, especially with obese patients over BMI 25. This is a randomized controlled trial comparing deep NMB with moderate NMB in laparoscopic subtotal gastrectomy in obese patients with gastric cancer. The design of the study is blinded (the surgical team and the research team are all blinded to the treatment); the attending anesthesiologist is not blinded. The primary endpoint is number of harvested lymph node that is critical point regarding quality of surgery in gastric cancer treatment. The secondary endpoint is intraoperative bleeding, surgeons' satisfaction.

The patients were randomly assigned to two groups using a computer-generated randomization table : 196 persons

* Deep neuromuscular block group (98persons)
* Moderate neuromuscular group (98persons) The patients are assigned to the deep NMB group or the moderate NMB group. The clinical research coordinator (CRC) uses a computer randomization program to determine the degree of muscle relaxation of each patient. Stratified block randomization is used to guarantee even distribution, which means that all participating hospitals are assigned moderate or deep NMB randomly in a 1:1 ratio. The CRC notifies the anesthesiologist of the degree of muscle relaxation just before the operation. Surgeons are blinded to the degree of muscle relaxation: They can enter the operating room after the muscle relaxation has been performed. A train-of-four (TOF) monitor is placed out of the surgeon's visual field. The anesthesiologist injects sugammadex after confirming the absence of the surgeon. The ward staff members who evaluate patient outcomes are blinded to the degree of muscle relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer patients with laparoscopic subtotal gastrectomy
* 19-75 years
* Body mass index(BMI) > 25kg/m2
* American Society of Anesthesiologists I-III

Exclusion Criteria:

* American Society of Anesthesiologists Class IV
* End stage renal disease (ESRD) patient
* Patients with allergy to muscle relaxants
* Patients with diseases that may affect muscle relaxation

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung soo Park, MD,PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Huh H, Choi SI, Kim JH, Jang YJ, Park JM, Kwon OK, Jung MR, Jeong O, Lee CM, Min JS, Kim JJ, An L, Yang KS, Park S, Lee IO; Deep Neuromuscular Block on Oncologic Quality of Laparoscopic Surgery in Obese Gastric Cancer Patients (DEBLOQS_GC) Study Group. Impact of the Deep Neuromuscular Block on Oncologic Quality of Laparoscopic Surgery in Obese Gastric Cancer Patients: A Randomized Clinical Trial. J Am Coll Surg. 2022 Mar 1;234(3):326-339. doi: 10.1097/XCS.0000000000000061. PMID 35213496
- [Derived] Lee Y, Ha D, An L, Jang YJ, Huh H, Lee CM, Kim YH, Kim JH, Park SH, Mok YJ, Lee IO, Kwon OK, Kwak KH, Min JS, Kim EJ, Choi SI, Yi JW, Jeong O, Jung MR, Bae HB, Park JM, Jung YH, Kim JJ, Kim DA, Park S. Comparison of oncological benefits of deep neuromuscular block in obese patients with gastric cancer (DEBLOQS_GC study): A study protocol for a double-blind, randomized controlled trial. Medicine (Baltimore). 2018 Dec;97(49):e13424. doi: 10.1097/MD.0000000000013424. PMID 30544421

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Neuromuscular Block Group: Sugammadex sodium 4mg/kg/IV after operation
  Sugammadex Sodium: 1. INDICATIONS AND USAGE BRIDION® is indicated for the reversal of neuromuscular blockade induced by rocuronium bromide and vecuronium bromide in adults undergoing surgery. BRIDION (sugammadex) injection is a sterile, clear, colorless to slightly yellow-brown, non-pyrogenic aqueous solution intended for intravenous infusion.
  2. DOSAGE AND ADMINISTRATION BRIDION (sugammadex) injection, for intravenous use, should be administered by trained healthcare providers familiar with the use, actions, characteristics, and complications of neuromuscular blocking agents (NMBA) and neuromuscular block reversal agents.
- Moderate Neuromuscular Group: Sugammadex sodium 2mg/kg/IV after operation
  Sugammadex Sodium: 1. INDICATIONS AND USAGE BRIDION® is indicated for the reversal of neuromuscular blockade induced by rocuronium bromide and vecuronium bromide in adults undergoing surgery. BRIDION (sugammadex) injection is a sterile, clear, colorless to slightly yellow-brown, non-pyrogenic aqueous solution intended for intravenous infusion.
  2. DOSAGE AND ADMINISTRATION BRIDION (sugammadex) injection, for intravenous use, should be administered by trained healthcare providers familiar with the use, actions, characteristics, and complications of neuromuscular blocking agents (NMBA) and neuromuscular block reversal agents.
Period: Overall Study
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
Started | 98 | 98
Completed | 88 | 93
Not Completed | 10 | 5
Not completed — Protocol Violation | 7 | 3
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Ten patients were excluded from the deep neuromuscular block group (7: protocol violation, 3: withdrew consent) and 5 patients were excluded from the moderate neuromuscular block group (3: protocol violation, 2: withdrew consent).
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group | Total
Number analyzed (Participants) | 88 | 93 | 181
Age, Categorical [Count of Participants; unit: Participants] — The effect of "Age" on oncological quality should be also considered. So, we categorize the patient according to "Age". Age is an important factor when considering phenotypic changes in health and disease. Age-related physiological changes can affect pharmacokinetics and pharmacodynamics of the drug. Typically, clinical trials categorize patients according to the age of 18 and 65 years.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 62 | 66 | 128
    >=65 years | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.6) | 60.0 (9.9) | 59.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — We tried to evaluate the impact of depth of neuromuscular block on oncological quality of laparoscopic surgery. In this circumstances, the effect of gender on oncological quality should be also evaluated. So, we categorize the patient according to "Sex".
  Participants
    Female | 60 | 62 | 122
    Male | 28 | 31 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 88 | 93 | 181
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: Body mass index (kg/m^2)] — Obesity hinders laparoscopic procedures and impedes oncological safety during laparoscopic cancer surgery. We aimed to evaluate whether deep neuromuscular block improves oncologic quality of laparoscopic cancer surgery in obese patients. So, we checekd wheter there is any difference in BMI between two groups.
  Body mass index (kg/m^2) | 27.6 (2.5) | 27.4 (2.1) | 27.5 (2.3)
ASA classification [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification offers clinicians a simple categorization of a patient's physiological status that can be helpful in predicting operative risk
  1. ASA I : No organic pathology or patients in whom the pathological process does not cause any systemic disturbance or abnormality.
  2. ASA II: moderate but definite systemic disturbance, caused by the condition that is to be treated or surgical intervention. (Mild diabetes, Anemia)
  3. ASA III: Severe systemic disturbance (Combinations of heart disease and respiratory disease)
  Participants
    ASA I | 14 | 8 | 22
    ASA II | 63 | 77 | 140
    ASA III | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Retrieved Lymph Nodes Per Participant
Description: Number of retrieved lymph nodes per participant, which was reported on final pathology report, after completing the laparoscopic surgery
Time Frame: within 14 days after operation
Population: This study originally intended to analyze whether a deeper depth of NMB can increase the number of retried LNs in obese gastric cancer patients. We tried to find a certain BMI point where the mean number of LNs showed a significant difference depending on the depth of NMB. BMI 28 was the starting point for the difference in the mean number of retrieved LNs.
Measure: Mean (Standard Deviation); unit: lymph nodes
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
Number analyzed (Participants) | 88 | 91
lymph nodes
  Total number of patients | 44.6 (17.5) | 41.5 (16.9)
  The patients with BMI ≥28kg/m^2: number analyzed (Participants) | 27 | 32
  The patients with BMI ≥28kg/m^2 | 49.2 (18.6) | 39.2 (13.3)

2. Secondary Outcome: Surgical Rating Score (SRS)
Description: Surgical rating score (SRS) at Four anatomical area during LN dissection
  During surgery, the surgeon reported the SRS based on the Leiden surgical rating scale (1=extremely poor, 2=poor, 3=acceptable, 4=good, 5=optimal) for each anatomical landmark (LN stations 4sb, 6, and 5 and the suprapancreatic area).
Time Frame: immediately after the operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
Number analyzed (Participants) | 88 | 91
score on a scale
  SRS in LN #4sb | 4.4 (0.9) | 4.3 (0.9)
  SRS in LN #5 | 4.2 (1.0) | 4.1 (1.0)
  SRS in LN #6 | 4.2 (0.9) | 4.2 (0.9)
  SRS in supra-pancreatic area | 4.1 (1.0) | 4.0 (1.1)
  Average SRS from 4 area | 4.2 (0.9) | 4.2 (0.9)

3. Secondary Outcome: Number of Participants With at Least One Interruption Event
Description: Interrupted event by patient movement, coughing, muscle spasm during operation
Time Frame: immediately after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
Number analyzed (Participants) | 88 | 91
Participants | 19 | 34

4. Secondary Outcome: Intraoperative Blood Loss Amount
Description: Amount of bleeding during operation
Time Frame: immediately after the operation
Measure: Median (Full Range); unit: mL
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
Number analyzed (Participants) | 88 | 91
mL | 77.5 [3.0 to 540.0] | 74.2 [3.0 to 500.0]

ADVERSE EVENTS:
Time Frame: Adverse event within 6 months were reported for every patients during outpatient clinic follow up.
Arm/Group | Deep Neuromuscular Block Group | Moderate Neuromuscular Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 0/98 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03196791/Prot_SAP_000.pdf